CLINICAL TRIAL: NCT04240990
Title: Development of a Diagnostic Prediction Score for Tuberculosis in Hospitalized Children With Severe Acute Malnutrition
Brief Title: Development of a Diagnostic Prediction Score for Tuberculosis in Hospitalized Children With Severe Acute Malnutrition (TB-Speed SAM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C18-28
Record Dates: First submitted 2019-10-24; First posted 2020-01-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis; Severe Acute Malnutrition
Keywords: Tuberculosis; Child; Malnutrition; Diagnosis; Screening
MeSH Terms: conditions — Tuberculosis; Severe Acute Malnutrition; Malnutrition; Disease | interventions — Algorithms; S-Adenosylmethionine

STUDY DESIGN:
Intervention Model Description: TB-Speed SAM is a multicentric, prospective diagnostic cohort study assessing several diagnostic tests that could result in the development of a score and algorithm for TB treatment decision in hospitalised children with SAM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort (Experimental): Children included in the cohort will all be in the same arm. The patients will benefit from standard-of-care TB diagnosis with additional diagnostic methods.
  Interventions: Other: Development of a score and algorithm for TB treatment decision in hospitalised children with SAM.

INTERVENTIONS:
Other: Development of a score and algorithm for TB treatment decision in hospitalised children with SAM. — The diagnostic strategy will include an initial clinical, radiographic and bacteriological evaluation of all enrolled children:
  * TB contact history
  * Suggestive TB symptoms in the previous 4 weeks
  * Physical examination
  * Clinical, anthropometric and biochemical assessment of malnutrition
  * Clinical assessment for other non-dietary causes of malnutrition
  * Digitalized CXR
  * Ultra performed on NPA and stool samples, and one gastric aspirate (GA)
  * Mycobacterial culture performed on two GAs
  * Abdominal ultrasonography
  * QuantiFERON®-TB Gold IGRA
  * Monocyte-to-Lymphocyte Ratio (MLR)
  * C-Reactive Protein (CRP)
  TB diagnosis will be made according to national TB guidelines.

SUMMARY:
TB-Speed SAM is a multicentric, prospective diagnostic cohort study conducted in two countries with high and very high TB incidence (Uganda and Zambia). It aims at assessing several diagnostic tests that could result in the development of a score and algorithm for TB treatment decision in hospitalised children with severe acute malnutrition (SAM).

DETAILED DESCRIPTION:
There is now strong evidence that undiagnosed and untreated TB increases the risk of death in children, especially those severely malnourished who are highly vulnerable. Specific decision-making tools are therefore urgently needed to guide clinicians from high TB burden and low-income countries to initiate treatment quickly in children with SAM with suspected TB.

A diagnostic prediction score and algorithm was recently proposed by the investigators for TB treatment decision in HIV-infected children with presumptive TB (developed in the ANRS 12229 PAANTHER 01 study). Based on easily collected clinical features, chest X-Ray (CXR), Xpert MTB/RIF, and abdominal ultrasonography, the score aims to help clinicians make a same-day treatment decision. Such a prediction score improving TB diagnosis and shortening time to treatment initiation would be a key benefit in children with SAM.

Based on this experience, the investigators are proposing a diagnostic cohort study enrolling hospitalized severely malnourished children. The study will include the evaluation of several diagnostic tests that could be integrated in the development of a prediction model and subsequent score for the diagnosis of TB in hospitalized children with SAM. This will include Xpert MTB/RIF Ultra performed on one nasopharyngeal aspirate (NPA) and one stool sample, CXR, Quantiferon (QFT) Interferon-Gamma Release Assay (IGRA), Monocyte-to-lymphocyte ratio (MLR), and ultrasonography, which has shown its interest for the diagnosis of TB in both HIV-infected adults and children. In the PAANTHER study, it detected abdominal lymphadenopathy in 50% of culture confirmed TB cases and 35% of all confirmed and unconfirmed cases, with a specificity of 85%.

Using logistic regression, a score will be developed for TB diagnosis, considering confirmed and unconfirmed TB as reference diagnosis, in hospitalized children with SAM. As a secondary objective, and in order to reduce costs, sample collection, and complexity of the diagnostic process, a first-step screening score (excluding Ultra, abdominal ultrasound, and CXR if possible) will be developed to identify children with presumptive TB who would benefit from further diagnostic testing.

Both scores will be internally validated using resampling and will be incorporated in a stepwise algorithm to guide practical implementation of the screening and diagnosis process. The stepwise algorithm will be discussed with local clinicians involved in the study to better adapt it for future use in their routine practice.

The study will be implemented at inpatient nutrition centres from three selected tertiary hospitals in Uganda, and Zambia. A total of 720 children <5 years old with WHO-defined severe acute malnutrition will be enrolled, that is approximately 240 participants per hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 59 months
* Severe acute malnutrition defined as weight-for-height Z score (WHZ) < -3 standard deviation (SD) or mid-upper arm circumference (MUAC) < 115 mm (in children over 6 months) or clinical signs of bilateral pitting oedema
* Hospitalized per hospital clinician's decision
* Parent/guardian informed consent

Exclusion Criteria:

- Ongoing TB treatment or history of intake of anti-TB drugs in the last 3 months

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 603 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the score obtained | 6 months
  Sensitivity of the score obtained using predicted probability cut-off with the prediction model for the diagnosis of TB, defined as either confirmed or unconfirmed using the updated Clinical Case Definition for Classification of Intrathoracic Tuberculosis
Specificity of the score obtained | 6 months
  Specificity of the score obtained using predicted probability cut-off with the prediction model for the diagnosis of TB

SECONDARY OUTCOMES:
Prevalence of TB among hospitalized children with SAM | 6 months
  Proportion of confirmed and unconfirmed TB in the study population
Clinical characteristics of TB disease in hospitalized children with SAM | 6 months
  Signs and symptoms of children with tuberculosis (confirmed and unconfirmed)
Bacteriological characteristics of TB disease in hospitalized children with SAM | 6 months
  Bacteriological characteristics (mycobacterial culture and drug susceptibility testing) of children with tuberculosis (confirmed and unconfirmed)
Biological characteristics of TB disease in hospitalized children with SAM | 6 months
  Haematological and immunological characteristics (full blood count, transaminases, CRP, IFN gamma) of children with tuberculosis (confirmed and unconfirmed)
Radiological characteristics of TB disease in hospitalized children with SAM | 6 months
  Radiological features (chest X-ray and abdominal US) of children with tuberculosis (confirmed and unconfirmed)
Sensitivity of the score obtained | 6 months
  Sensitivity of the score obtained using predicted probability cut-off with the screening prediction model for the identification of children with presumptive TB requiring further diagnostic evaluation
Specificity of the score obtained | 6 months
  Specificity of the score obtained using predicted probability cut-off with the screening prediction model for the identification of children with presumptive TB requiring further diagnostic evaluation
Estimated time to TB treatment decision in hospitalized children with SAM | 6 months
  Estimated time to TB treatment decision in hospitalized children with SAM, with and without presumptive TB based on the first-step screening prediction score
Diagnostic accuracy measures: 1/ Sensitivity of the different tests evaluated for the diagnosis of TB | 6 months
  Sensitivity of the different tests evaluated for the diagnosis of TB (Ultra performed on NPA and stools, CXR, abdominal ultrasound, QFT, MLR, CRP)
Diagnostic accuracy measures: 2/ Specificity of the different tests evaluated for the diagnosis of TB | 6 months
  Specificity of the different tests evaluated for the diagnosis of TB (Ultra performed on NPA and stools, CXR, abdominal ultrasound, QFT, MLR, CRP)
Diagnostic accuracy measures: 3/ Negative predictive value of the different tests evaluated for the diagnosis of TB | 6 months
  Negative predictive value of the different tests evaluated for the diagnosis of TB (Ultra performed on NPA and stools, CXR, abdominal ultrasound, QFT, MLR, CRP)
Diagnostic accuracy measures: 4/ Positive predictive value of the different tests evaluated for the diagnosis of TB | 6 months
  Positive predictive value of the different tests evaluated for the diagnosis of TB (Ultra performed on NPA and stools, CXR, abdominal ultrasound, QFT, MLR, CRP)
Diagnostic accuracy measures: 5/ AUROC of diagnostic prediction models with and without the different tests results | 6 months
  Area Under the Receiver Operating Characteristics curve
Diagnostic accuracy of Ultra performed on one NPA and one stool sample against a specific microbiological reference standard including Ultra and mycobacterial culture from gastric aspirates | 6 months
  Proportion of NPAs and stool samples with mycobacterium tuberculosis detected using Ultra
Proportion of children with NPA and stool samples collected as per study protocol | 6 months
  Feasibility of NPA and stool samples collection defined as the proportion of children with NPA and stool samples collected as per study protocol
Proportion of NPA-related adverse events (AEs) | 6 months
  Safety of NPA collection defined as proportion of AEs (vomiting, nose bleeding, low oxygen saturation, respiratory distress) occurring during NPA
Tolerability of NPA collection: 1/ Discomfort/pain/distress experienced by the child as assessed by the child | Within 3 days of inclusion
  Discomfort/pain/distress experienced by the child during NPA collection, as assessed by the child using the Wong-Baker face scale (in a subset of children).
  Scale range: 0 (no hurt) - 5 (hurts worst)
Tolerability of NPA collection: 2/ Discomfort/pain/distress experienced by the child as assessed by the parents | Within 3 days of inclusion
  Discomfort/pain/distress experienced by the child during NPA collection, as assessed by the parents using the visual analog scale (in a subset of children).
  Scale range: 0 (no pain) - 10 (pain as bad as it could possibly be)
Tolerability of NPA collection: 3/ Discomfort/pain/distress experienced by the child as assessed by the nurse | Within 3 days of inclusion
  Discomfort/pain/distress experienced by the child during NPA collection, as assessed by the nurses using the "Face Legs Activity Cry Consolability" behavioral pain scale (in a subset of children).
  Total score range: 0 (relaxed and comfortable) - 10 (severe discomfort/pain). Each item of the FLACC scale - Face, Legs, Activity, Cry, Consolability - has 3 possible quotes: 0 or 1 or 2, with a precise description provided to help with the rating. The total score is obtained by adding individual item scores.
Mortality at 6 months | 6 months
  Mortality at 6 months in children with SAM, with or without TB treatment
Percentage weight gain 6 months | 6 months
  Weight gain and WHZ at 6 months in children with SAM, with or without anti-TB treatment
TB treatment outcomes | 6 months
  TB treatment outcomes as defined per WHO guidelines (Cured, Treatment completed, Treatment failed, Died, Lost to follow-up, Not evaluated, Treatment success)

OTHER OUTCOMES:
Incremental cost-effectiveness ratio (ICER) | 32 months
  Incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marcy, MD, PhD, Principal Investigator — University of Bordeaux, France; Maryline Bonnet, MD, PhD, Principal Investigator — Institut de Recherche pour le Développemnt (IRD) Montpellier, France; Eric Wobudeya, MD, PhD, Principal Investigator — MU-JHU Care Ltd, Kampala, Uganda
Locations (3):
- Mulago National Referral Hospital, Kampala, Uganda
- Zambia (2):
  - Lusaka University Teaching Hospital, Lusaka
  - Arthur Davidson Children Hospital, Ndola

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chabala C, Roucher C, Ton Nu Nguyet MH, Babirekere E, Inambao M, Businge G, Kapula C, Shankalala P, Nduna B, Mulenga V, Graham S, Wobudeya E, Bonnet M, Marcy O; TB-Speed SAM study group. Development of tuberculosis treatment decision algorithms in children below 5 years hospitalised with severe acute malnutrition in Zambia and Uganda: a prospective diagnostic cohort study. EClinicalMedicine. 2024 Jun 20;73:102688. doi: 10.1016/j.eclinm.2024.102688. eCollection 2024 Jul. PMID 39007063
- [Result] d'Elbee M, Mafirakureva N, Chabala C, Huyen Ton Nu Nguyet M, Harker M, Roucher C, Businge G, Shankalala P, Nduna B, Mulenga V, Bonnet M, Wobudeya E, Marcy O, Dodd PJ. Treatment decision algorithms for tuberculosis screening and diagnosis in children below 5 years hospitalised with severe acute malnutrition: a cost-effectiveness analysis. EClinicalMedicine. 2025 Apr 19;83:103206. doi: 10.1016/j.eclinm.2025.103206. eCollection 2025 May. PMID 40291345
- See also: TB-Speed project official website — http://www.tb-speed.com